CLINICAL TRIAL: NCT02715596
Title: Relationship Between Changes in Body Composition and Supplementation With EPA in Patients Diagnosed With Squamous Cell Carcinoma of Head and Neck Locally Advanced (Stage III-IVb)
Brief Title: Changes in Body Composition After EPA Supplementation in Head and Neck Patients
Acronym: hepaneck
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Català d'Oncologia (Other)
Collaborators: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PR 261/14
Record Dates: First submitted 2015-02-12; First posted 2016-03-22 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: head and neck; eicosapentanoic acid; body composition
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: eicosapentanoic acid (EPA) versus placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo (EPA)
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention A (Experimental): 2.7 g EPA supplementation in a 15 cc emulsion stick-pack
  Interventions: Dietary Supplement: EPA supplementation
- Intervention B (Placebo Comparator): Placebo supplementation in a 15 cc emulsion stick-pack
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: EPA supplementation — 2.7 g EPA supplementation in a 15 cc emulsion stick-pack
  Arms: Intervention A
Other: Placebo — placebo in 15 cc emulsion stick-pack
  Arms: Intervention B

SUMMARY:
Evaluates the effect of EPA supplementation in terms of muscle mass in patients with squamous cell carcinoma of the head and neck locally advanced

DETAILED DESCRIPTION:
This study is designed to evaluate the effect of EPA supplementation on muscle mass in patients with squamous cell carcinoma of the head and neck locally advanced (stage III-IVb) to assess that supplementation with EPA can maintain muscle mass along the oncologic treatment. Other aims are to evaluate the nutritional status, acute and chronic toxicities related with the loss of muscle mass and the impact of the EPA supplementation on overall and disease-free survival.

ELIGIBILITY:
Inclusion Criteria:

* - Age between 18 and 75 years inclusive.
* A performance status 0-1 according to ECOG (Eastern Cooperative Oncology Group) scale at the time of inclusion in the study.
* Expectancy greater than 3 months life.
* Location: oral cavity, oropharynx, larynx,hypopharynx, nasopharynx and sinuses.
* Patients with squamous cell carcinoma of the head and neck classified as locally advanced (Stage III, IVa-IVb).
* Patients with medical conditions to receive neoadjuvant chemotherapy (CT) induction followed by radiotherapy (RDT) normo fraction combined with QT or biological.
* Neutrophil ≥1500 / mm3, platelet count ≥150,000 / mm3 and hemoglobin ≥10g / dL.
* Adequate liver function: total bilirubin ≤ 1 x ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN; Alkaline phosphatase (ALP) ≤ 5 x ULN.
* Serum albumin-adjusted calcium ≤ 1.25 x upper limit of normal (ULN).
* Using an effective contraceptive method for patients of both sexes where the risk of conception and / or pregnancy.
* Signature of written informed consent before any study-specific procedures

Exclusion Criteria:

* - Metastatic disease (stage IVc).
* Surgery, radiotherapy and / or chemotherapy prior to study disease treatment.
* T3 N0-1 larynx.
* Other stadiums than III or IV without distant metastases and stable disease.
* Another synchronous squamous carcinoma.
* Diagnosis of other malignancy within the past 5 years, except in situ of the cervix and / or adequately treated basal cell carcinoma skin cancer.
* Active infection (infection requiring intravenous antibiotic), including active tuberculosis and HIV diagnosed.
* Uncontrolled hypertension defined as systolic blood pressure ≥180mm Hg and / or diastolic blood pressure≥ 130 mm Hg at rest.
* Pregnancy (absence must be confirmed with β-HCG (Human chorionic gonadotropin) serum test) or lactating.
* Systemic, chronic immune and concomitant treatment, or hormonal treatment of cancer.
* Other concomitant antineoplastic treatment.
* Clinically significant coronary artery or a history of myocardial infarction in the last 12 months or high risk of uncontrolled arrhythmia or uncontrolled heart failure.
* Chronic obstructive pulmonary disease that would have required ≥3 hospitalizations in the last 12 months.
* Uncontrolled active peptic ulcer.
* Presence of a psychological or medical illness that prevented the study by the patient or to grant the signature on the informed consent.
* Abuse of known drugs (with the exception of heavy drinking).
* Allergic reaction known against any component of study treatment.
* Previous treatment with monoclonal antibodies or other inhibitors of signal transduction or treatment directed against the EGFR (epidermal growth factor receptor).
* Any experimental therapy within 30 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
The effect of supplementation with EPA on muscle mass during a conservative non-surgical treatment of organ in patients with squamous cell carcinoma of head and neck locally advanced. | 3 years
  To evaluate the effect of supplementation with EPA on muscle mass during a conservative non-surgical treatment of organ in patients with squamous cell carcinoma of head and neck locally advanced.

SECONDARY OUTCOMES:
the effect of supplementation with EPA on muscle mass after induction chemotherapy using imaging such as CT scan | 10 weeks
  To evaluate on muscle mass using imaging such as CT scan
Evolution of nutritional status of patients over oncology-specific treatment in both arms. using PG-VGS | 1 year
  To assess the evolution of nutritional status using PG-VGS (patient generated subjective global assessment)
The effect of supplementation with EPA regarding acute toxicity during treatment.using the CTCAE v4 criteria | 1 year
  To evaluate the frequency of acute toxicity using the CTCAE v4 criteria
The effect of supplementation with EPA in relation to chronic toxicity 2 years after oncologic treatment. (using the CTCAE v4 criteria) | 2 years
  To evaluate the frequency of chronic toxicity using the CTCAE v4 criteria
The impact of supplementation with EPA in the loco-regional control at 2 years after completing cancer treatment. | 2 years
  To evaluate whether the effect of supplementation with EPA influences the loco-regional control using a CT scan
The effect of supplementation with EPA on the perceptions of patients through quality of life validated questionnaires. | 2 year
  o To evaluate and compare the effect of supplementation with EPA on the perceptions of patients through quality of life questionnaires (QLQ) validated such as QLA-C30
The adherence to EPA. (using record EPA/placebo dispensing and return and blood samples at baseline and throughout the cancer treatment) | 1 year
  To assess adherence to EPA using record EPA/placebo dispensing and return and blood samples at baseline and throughout the cancer treatment of the EPA concentration in the erythrocyte membrane
The functional status of patients throughout the treatment. (functional status using hand grip) | 1 year
  To evaluate the functional status using hand grip
The need for nutritional support and nutritional intervention required during cancer treatment among patients supplemented with EPA or placebo. | 1 year
  To compare the need for nutritional support and nutritional intervention required using data collection sheet with the different types of nutritional support, days of each nutritional intervention and adherence to it.
The impact of supplementation with EPA on the recurrence-free survival at 2 years after completing cancer treatment. | 2 years
  To evaluate whether the effect of supplementation with EPA influences the recurrence-free survival using a CT scan
The impact of supplementation with EPA on the overall survival at 2 years after completing cancer treatment. | 2 years
  To evaluate whether the effect of supplementation with EPA influences the overall survival using a CT scan
The effect of supplementation with EPA on the perceptions of patients through quality of life validated questionnaires. | 2 years
  To evaluate and compare the effect of supplementation with EPA on the perceptions of patients through quality of life questionnaires (QLQ) validated such as QLQ-H&N35
The functional status of patients throughout the treatment. (functional status using performance status scale) | 1 year
  To evaluate the functional status using performance status scale

CONTACTS AND LOCATIONS:
Overall Officials: Lorena Arribas, RD, MsC, Principal Investigator — Institut Català d'Oncologia
Locations (1):
- Institut Catala d'Oncologia- L'Hospitalet, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes